CLINICAL TRIAL: NCT01364493
Title: An Open-label, Single Arm Study to Evaluate the Efficacy and Safety of Trastuzumab in Combination With Capecitabine and Oxaliplatin (XELOX) as a First-line Chemotherapy for Inoperable, Locally Advanced or Recurrent and/or Metastatic Gastric Cancer
Brief Title: A Study to Evaluate the Efficacy and Safety of Trastuzumab in Combination With Capecitabine and Oxaliplatin as First-line Chemotherapy for Inoperable, Locally Advanced or Recurrent and/or Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, M.D., Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGOG1001
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Gastric Cancer
Keywords: HER2-positive; adenocarcinoma of the stomach or gastro-esophageal junction; Inoperable; locally advanced; recurrent; metastatic
MeSH Terms: conditions — Stomach Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Trastuzumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trastuzumab+Capecitabine+Oxaliplatin (Experimental): Trastuzumab will be administered at a loading dose of 8 mg/kg (on day 1) followed by 6mg/kg i.v. infusion every 3 weeks.
  Capecitabine 2000mg/m2d, d1-14; q3w, Oxaliplatin 130mg/m2 d1; q3w, 6 cycles
  Interventions: Drug: Trastuzumab+Capecitabine+Oxaliplatin

INTERVENTIONS:
Drug: Trastuzumab+Capecitabine+Oxaliplatin — Trastuzumab will be administered at a loading dose of 8 mg/kg (on day 1) followed by 6mg/kg i.v. infusion every 3 weeks.
  Capecitabine 2000mg/m2d, d1-14; q3w, Trastuzumab and capecitabine are to be continued until disease progression or intolerable toxicity.
  Oxaliplatin 130mg/m2 d1; q3w, 6 cycles
  Other Names: Herceptin; Xeloda; Eloxatin

SUMMARY:
Although the overall incidence of gastric cancer has steadily declined in many Western countries during the last few decades, it is still one of the most common tumors in China. It is now well recognised that combination chemotherapy regimens improve patient outcomes, but there is no accepted global standard regimen for advanced gastric cancer.

The ToGA study was the first randomized, prospective, multicenter, phase III trial to show the efficacy and safety of Trastuzumab in HER2- positive GC. Trastuzumab reduced the risk of death by 26% (HR 0.74; 95% CI 0∙60, 0∙91; p=0∙0046) when combined with a reference chemotherapy (Capecitabine plus Cisplatin) and prolonged the median survival by nearly 3 months (from 11.1 to 13.8 months) in patients with HER2-positive(FISH+ or IHC3+) advanced GC.

Oxaliplatin has been shown to be as effective as cisplatin, and exhibits a favorable toxicity profile with a substantially lower rate of nephrotoxicity, ototoxicity, and myelosuppression.

In the current study, the efficacy and safety of Trastuzumab in combination with Oxaliplatin/capecitabine chemotherapy will be evaluated in Chinese patients with HER2 positive advanced or recurrent gastric cancer.

DETAILED DESCRIPTION:
Trastuzumab will be administered at a loading dose of 8 mg/kg (on day 1) followed by 6mg/kg i.v. infusion every 3 weeks.

Trastuzumab is to be continued until disease progression or intolerable toxicity.

Capecitabine (Xeloda) 2000mg/m2d, d1-14; q3w, until disease progression or intolerable toxicity.

Oxaliplatin 130mg/m2 d1; q3w, 6 cycles

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the stomach or gastro-oesophageal junction with inoperable locally advanced or recurrent and/or metastatic disease, not amenable to curative therapy.
2. Measurable disease, according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.0), assessed using imaging techniques (CT or MRI).
3. HER2 positive tumour (primary tumour or metastasis) as assessed by the central laboratory. (Both IHC and Dual SISH will be performed on all patients in the central laboratory.)
4. ECOG Performance status 0, 1 or 2.
5. Life expectancy of at least 3 months.
6. Male or female. Age ≥ 18 years.
7. Signed informed consent.

Exclusion Criteria:

1. Previous chemotherapy for advanced/metastatic disease (prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrolment into the study; the total dose of cisplatin should be less than 300mg/m2, adjuvant/neoadjuvant therapy with oxaplatin is not allowed).
2. No prior use of EGFR-targeting drugs,such as Trastuzumab,lapatinib or other TKIs.
3. Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome (e.g. patients with partial or total gastrectomy can enter the study, but not those with a jejunostomy probe).
4. Patients with active (significant or uncontrolled) gastrointestinal bleeding.
5. Residual relevant toxicity resulting from previous therapy (with the exception of alopecia), e.g. neurological toxicity ≥ grade 2 NCI-CTCAE 4.0.
6. Other malignancy within the last 5 years, except for carcinoma in situ of the cervix, or basal cell carcinoma.
7. Neutrophil count < 1.5 × 109/L, or hemoglobin < 90 g/L,or platelet count < 100 × 109/L.
8. Serum bilirubin > 1.5 × upper limit of normal (ULN); or, AST or ALT > 2.5 × ULN(or > 5 × ULN in patients with liver metastases); or, alkaline phosphatase > 2.5 × ULN (or > 5 × ULN in patients with liver metastases, or > 10 × ULN in patients with bone but no liver metastases); or, albumin < 25 g/L.
9. Creatinine clearance < 60 mL/min.
10. History of documented congestive heart failure; angina pectoris requiring medication;evidence of transmural myocardial infarction on ECG; poorly controlled hypertension (systolic BP > 180 mmHg or diastolic BP > 100 mmHg); clinically significant valvular heart disease; or high risk uncontrollable arrhythmias.
11. Baseline LVEF < 50% (measured by echocardiography or MUGA).
12. Patients with dyspnoea at rest due to complications of advanced malignancy or other disease, or who require supportive oxygen therapy.
13. Patients receiving chronic or high dose corticosteroid therapy. (Inhaled steroids and short courses of oral steroids for anti-emesis or as an appetite stimulant are allowed).
14. Clinically significant hearing abnormality.
15. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
16. History or clinical evidence of brain metastases.
17. Serious uncontrolled systemic intercurrent illness, e.g. infections or poorly controlled diabetes.
18. Positive serum pregnancy test in women of childbearing potential.
19. Subjects with reproductive potential not willing to use an effective method of contraception.
20. Received any investigational drug treatment within 4 weeks of start of study treatment.
21. Radiotherapy within 4 weeks of start of study treatment (2 week interval allowed if palliative radiotherapy given to bone metastastic site peripherally and patient recovered from any acute toxicity;prior adjuvant radiotherapy is allowed if complete at least 6 months ).
22. Major surgery within 4 weeks of start of study treatment, without complete recovery.
23. Patients with known active infection with HIV, HBV, or HCV.
24. Known hypersensitivity to any of the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 6 -8 weeks
  CT/MRI will be performed every 2 cycles of treatment for efficacy evaluation

SECONDARY OUTCOMES:
progression free survival | 1 year
  the follow-up visit of PFS will be performed every 6 weeks
overall survival of participants | 2 years
  OS means that from the first dose of treatment drug to death or lost, the follow-up visit will be performed every 3 months till death or lost
adverse events | during the treatment in the hosptital,an expected average of 3 weeks
  participants will be followed for the duration of hospital stay, an expected average of 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Lin Shen, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Gong J, Liu T, Fan Q, Bai L, Bi F, Qin S, Wang J, Xu N, Cheng Y, Bai Y, Liu W, Wang L, Shen L. Optimal regimen of trastuzumab in combination with oxaliplatin/ capecitabine in first-line treatment of HER2-positive advanced gastric cancer (CGOG1001): a multicenter, phase II trial. BMC Cancer. 2016 Feb 8;16:68. doi: 10.1186/s12885-016-2092-9. PMID 26857702